CLINICAL TRIAL: NCT04179903
Title: Efficacy and Safety of the Exercise Program in Women With Post-menopausal Osteoporosis: Randomized Trial Comparing Gym Versus Home Training
Brief Title: Efficacy and Safety of the Physical Activity Program in Women With Post-menopausal Osteoporosis
Acronym: ACTLIFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 45/18
Record Dates: First submitted 2019-06-04; First posted 2019-11-27 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Osteoporosis, Postmenopausal; Physical Activity
Keywords: osteoporosis; Gym Training; physical activity; home training
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Motor Activity; Osteoporosis | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gym Trainer (Active Comparator): Physical Activity program is performed in a group in a gym (Gym Group Training-GGT), with activity sessions conducted by a trainer graduated in Science and Techniques of Preventive and Adapted Physical Activity
  Interventions: Other: Physical activity
- Individual Home (Active Comparator): Physical Activity program is performed at home individually (Individual Home Training-IHT), without the supervision of a trainer during the exercise session.
  Interventions: Other: Physical activity

INTERVENTIONS:
Other: Physical activity — Physical Activity program is performed in a group in a gym and at home

SUMMARY:
The study will be single blinded since professionals who will evaluate patients will not know to which exercise group patients have been assigned.

The investigators hypothesize that effectiveness and safety of the exercise program are equal when administered as gym trainer or individual home trainer. However, the investigators expect differences in adherence among the two groups which may cause different impact on the outcome measures.

Given the large amount of evidence on the efficacy of Physical Activity in women with Osteoporosis, the investigators considered it ethically unacceptable to advise a control group inactivity. On the other hand, it seemed particularly relevant for the purpose of addressing the advice to the improvement of the active lifestyle, to evaluate the impact of the ACTLIFE exercise program when administered as gym trainer or individual home trainer

DETAILED DESCRIPTION:
The present study is carried out within the project "Physical ACTivity: the tool to improve the quality of LIFE in osteoporosis people" (ACTLIFE) and is funded within the Erasmus Plus Sport program (Grant Agreement N2017-2128/001-001).

It is aimed at evaluating differences in efficacy and safety of a PA program specifically designed for improving physical function and, here in after, QoL in post menopausal women with Osteoporosis (T-score <-2,5) under usual pharmacological treatment, when administered as gyms as group training (GGT) or Individual Home Training IHT. During the study patients will be recommended to maintain their usual pharmacological treatment for OP, as prescribed.

The primary objective of the study is to compare modifications of QoL measured with the Short Osteoporosis Quality of Life Questionnaire (ECOS-16) induced by the ACTLIFE exercise programme when administered as IHT or GGT. ECOS-16 is a specific-disease instrument with the purpose to measure the health related QoL (HRQoL) in post menopausal women with OP.

The secondary objectives of the study are to investigate differences between IHT and GGT on domains which are considered to be determinants of QoL:

* WHO Disability Assessment Schedule (WHODAS) which evaluates the six activity and participation domains of the International Classification of Functioning, Disability and Health (ICF): cognition, mobility, self-care, interacting with other people, life activities, participation.
* Fear of falls evaluated by the Falls Efficacy Scale International (FES-I);
* Walking (6-Minute Walk Test), standing balance (stability Index), muscle force (hand grip), postural alignment (occiput-wall distance) and joint mobility will be also evaluated as fundamental prerequisites of motor behavior;
* Body Mass index and body composition.

The adherence of each patient to the exercise program will be monitored. The adherence will be measured as percent of exercise sessions actually performed /total number of scheduled exercise sessions. The investigators hypothesize that effectiveness and safety of the exercise program are equal when administered as GGT or IHT. However, the investigators expect differences in adherence among the two groups which may cause different impact on the outcome measures. In the context of the evaluation of adherence to the program, the satisfaction of the participants for the ACTLIFE program administered as GGT or IHT at the end of the 12 months of exercise will be evaluated with a specific questionnaire based on 7-point Likert scale and the reasons of abandoning the exercise program (question with structured answers). Education attainment, work activity, marital status and home-gym distance will be also recorded since recognized to influence the adherence in an exercise program.

The ultimate goal of the ACTLIFE exercise program is to increase physical activity in a sedentary population. The exercise program, through its beneficial effects on health, is expected to generate a virtuous circle of greater activity and participation. In this context, to evaluate differences between GGT or IHT, the investigators introduced in the study protocol the Physical Activity Scale for the Elderly (PASE). PASE is an easily scored survey designed specifically to measure the weekly physical activity in adult and aged population. Its score combines information on leisure, household and occupational activity.

RT with two parallel groups: in the first group the 12-month ACTLIFE program is performed as IHT, while in the second as GGT. The study will be single blinded since professionals who will evaluate patients will not know to which exercise group they have been assigned. Patients will be assessed at baseline and after 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* post menopausal women aged >40 years (with or without history of fractures, with or without pharmacological therapy for OP)
* lumbar spine or femur T-score ≤-2,5
* functional motor capacity normal or moderately reduced (Short Physical Performance Battery)
* sedentary life style (having exercised less than 30 minutes per week in the last 6 months).

Exclusion Criteria are:

* secondary OP49, impairment of communicative and/or sensorial functions so severe to make impossible understanding or executing trainer's instructions (dementia, aphasia, blindness, deafness);
* heart failure (NYHA class >2);
* unstable angina, pulmonary disease requiring oxygen therapy;
* symptomatic peripheral arteriopathy;
* myocardial infarction or hospital admission in the previous 6 months,
* symptomatic orthostatic hypotension;
* hypertension in poor pharmacologic control (diastolic >95 mmHg, systolic >160 mmHg),
* previous implant of prosthesis at upper or lower limbs,
* relevant neurological condition impairing motor or cognitive function, any other condition that the medical doctor (MD) considers to contraindicate the participation in an exercise program of moderate intensity.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Quality of life questionnaire | 12 months
  Assessment of health related quality of life in osteoporosis - ECOS-16 questionnaire measures the HRQoL in postmenopausal women with osteoporosis. The 16 items are divided into 4 dimensions.
  The score of each item ranges from 1 to 5. A single summary score obtained from the arithmetic mean of the answered items, so the total score ranges from 1 (best HRQoL) to 5 (worst HRQoL).

SECONDARY OUTCOMES:
Disability | 12 months
  WHODAS has six domains of life
  1. Cognition understanding and communicating
  2. Mobility
  3. Self-care
  4. Getting along
  5. Life activities Summing of recorded item scores within each domain after the converting the summary score into a metric raging from 0 to 100 ( 0 = no disability - 100 = full disability)
Fear of falls | 12 months
  Falls Efficacy Scale International - FES-I The score contains 16 items scored on a four point scale (1= not all concerned to 4= very concerned
  To calculate the FES-I or Short FES-I score when all items are completed, simply add the scores for each item together to give a total that ranges as follows:
  Minimum 16 (no concern about falling) to maximum 64 (severe concern about falling)
Walking | 12 months
  6-Minute Walk Test The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance (m) covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
  An increase in the distance walked indicates improvement in basic mobility.
standing balance | 12 months
  Standing balance will be estimated by the validated Stability Index for both right and left lower limb.
  It evaluates proprioceptive control, visual dependence, and the risk of fall and injury.
  The Stability Index is a score (0-100 %). 100% is high
Muscle force | 12 months
  Hand grip (KG)
joint mobility | 12 months
  Hip range of motion in degree, knee range of motion in degree, shoulder range of motion in degree
Body Mass Index | 12 months
  Weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Ripamonti, Principal Investigator — IOR
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No